CLINICAL TRIAL: NCT02414529
Title: Efficacy of Vitamin D Therapy on Glucose Homeostasis in Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 12-03213
Record Dates: First submitted 2015-04-01; First posted 2015-04-10 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Ergocalciferols; Vitamin D

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo group (Placebo Comparator): Placebo group B: single blinded to patients, receive 6 capsule PO (placebo) at once.
  Subjects are blinded then they will crossover groups
  Interventions: Drug: Placebo
- Treatment group (Active Comparator): Group A will receive 6 capsules (50.000 units/each) of vitamin D2(ergocalciferol) at once.
  Subjects are blinded then they will crossover groups.
  Interventions: Drug: Vitamin D2

INTERVENTIONS:
Drug: Vitamin D2 — Ergocalciferol 5000 units capsules given. 300,000 units PO once.
  Other Names: ergocalciferol, Vitamin D
  Arms: Treatment group
Drug: Placebo
  Arms: Placebo group

SUMMARY:
The purpose of this study is to see whether giving a Vitamin D supplement to vitamin D deficient obese children and adolescents will decrease the risk of getting diabetes (Disease in which the person has high blood sugar).

The number of vitamin D deficiency in U.S. children and teenagers has grown dramatically over the past 30 years. There are some reports suggesting that vitamin D supplementation in adults with pre diabetes (blood glucose higher than normal) and vitamin D treatment will prevent diabetes.

DETAILED DESCRIPTION:
Participation will involve 3 visits (6 weeks apart) to the Clinical and Translational Science Institute (CTSI), which should happen 2-3 weeks after you have consented to participate in this study. The total duration of the study and the time you/your child will spend in the CTSI will be 2.5 hours for each visit.

Number of adolescents/children will enroll in this study:20.

Visit 1 A doctor will perform a complete physical examination. The child will have his/her weight and height measured .Blood pressure and vital signs will check each visit.

Of the 2 hours spent in the hospital, 1/2 hour is allocated to getting measurements, weight, and vitals and putting in an intravenous line and drawing fasting labs. The oral glucose tolerance test will take about 2 hours. To test for insulin sensitivity (Risk marker of Diabetes), oral Glucose Tolerance Test (OGTT) will be done. OGTT is used to diagnose Diabetes and Pre Diabetes. The child will first have blood samples drawn, and then will drink oral glucose soda. Blood samples will be obtained over 2 hours. A total of 5-7 teaspoons, which is 25-35 cc of blood will be taken during this test. Of this 15 cc will be drawn during the OGTT. A doctor or nurse will be monitoring the child throughout the test. If he/she develops low blood sugar, they will be treated appropriately with glucose.

Blood samples obtained at the start of the OGTT will be used to measure various markers of insulin sensitivity, vitamin D level and marker of bone health as vitamin D deficiency can causebone loss. This blood will be stored in the CTSI core laboratory in the CTSI for duration of this study. The blood samples will be stored without child's name or any other identifying information on them. The samples will be destroyed once the study is completed.

After the OGTT done, your child will receive a one time high dose of vitamin D (group A) or placebo (capsule containing no medication) (Group B). This way of treating of low vitamin D levels with one time high dose of vitamin D is safe and has been studied in adolescents.

The child has 50/50 chance to be in either group. Neither he/she nor you will know if he/she is getting Vit D or placebo. At week 7, your child needs to return to CTSI for 2nd study for physical check-up, blood test and urine test using the same method as the 1st visit. The urine testing will be done to test for urinary calcium as this could be a sign of vitamin D toxicity.

After the 2nd study done, your child will be reassigned to alternate treatment group and will receive either vitamin D or placebo. That means that if he/she was getting a placebo at the first visit then he/she will get a real Vit D this time. If he/she was getting vit D at the first visit, he/she will get a placebo at this visit.

At week 12 after completion of the 2nd course of medication, you and your child will have to come back for the final blood and urine study using the same method as the first and 2nd study.

At this your child will have an oral glucose tolerance test, blood and urine tests. The urine testing will be done to test for urinary calcium as this could be a sign of vitamin D toxicity. If your child has high urine calcium he/she will not be allowed to participate in the study We guarantee that your child will receive the treatment for lack of vitamin D either the first half or latter half of the study. However, you will not know what medication your child will receive during the entire study. We will set an appointment to see us in 2weeks at the Endocrine clinic; however, it will be not part of the study. We will go over the results of the study at that time and will see if any further treatment with Vitamin D is required for your adolescent.

You and your child will have to come back to CTSI at the end of week 12 for post-therapy study. After a minimum 10-hour fast, participants will come to the CTSI, during which your child will have his/her weight and height measured. Blood Pressure will be measured. Post vitamin D therapy OGTT. Vitamin D level and markers for bone health will again be measured using same method as day 1. Urine will be collected for urinary calcium level, using same method as day 1.

ELIGIBILITY:
Inclusion Criteria:

1. Obese subjects - BMI at or above the 95th percentile for children of the same age and sex. Only obese subjects will be selected given that they are the highest risk group of developing insulin resistance and Type II Diabetes and therefore with be most likely to demonstrate glucose pertubation.
2. Pubertal: Testicular volume ≥ 6 ml Prader (M) and Tanner III breast development or greater (F)
3. 12- 18 years regardless of gender, race or economic circumstance
4. Pre diabetes/high risk of diabetes using criteria of HbA1C between 5.7 - 6.4% as defined by the American Diabetes Association (ADA)
5. 25-OH vitamin D level less than 20 ng/ml (50 nmol/liter)
6. Subjects must be willing to comply with study protocol requirements

Exclusion Criteria:

1. Treatment on medication known to effect vitamin D, calcium and glucose metabolism, such as glucocorticoids, thiazolidinediones, metformin, anticonvulsants metabolized through cytochrome P-450 (phenytoin, carbamazepine, phenobarbital, sodium valproate).
2. Subjects will be excluded from the study if they have taken any form of vitamin D supplementation greater than 400 IU daily in the preceding 3 months.
3. Significant major organ system illness
4. History of nephrolithiasis or hypercalcemia
5. Females who are pregnant
6. Significant psychiatric illness: schizophrenia, bipolar disorder, active substance abuse, and uncontrolled major depression.
7. Attendance at tanning salon

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Whole Body Insulin Sensitivity (WBISI) | 18 weeks
  measured by the OGTT
Insulinogenic index | 18 weeks
  meassured by OGT

SECONDARY OUTCOMES:
Vitamin D 25 OH | 18 weeks
  pre and post treatment changes in serum vitamin D 25 OH.
PTH level | 18 weeks
  changes in the level PTH pre and post treatment
Vitamin D toxicity | 18 weeks
  will measure metabolic profile to monitor toxicity such us: calcium level in serum and urine, phosphate, vitamin D

CONTACTS AND LOCATIONS:
Overall Officials: Preneet Brar, Principal Investigator — NYU School of Medicine
Locations (1):
- bellevue hospital CTSI, New York, New York, United States